CLINICAL TRIAL: NCT05492968
Title: The Effect of Epinephrine, Norepinephrine and Phenylephrine on Intraoperative Hemodynamic Performance - a Prospective Double-blinded Randomized Clinical Trial
Brief Title: The Effect of Epinephrine, Norepinephrine and Phenylephrine on Intraoperative Hemodynamic Performance
Acronym: RACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RACE_01
Record Dates: First submitted 2022-07-28; First posted 2022-08-09 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Output, Low; Cardiac Output, High; Perfusion; Complications
Keywords: Norepinephrine; Epinephrine; Phenylephrine; Major abdominal surgery; Intraoperative Cardiac Output; Intraoperative Hemodynamic; Intraoperative Perfusion
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High | interventions — Epinephrine; Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Epinephrine Group (Experimental): Patients in the epinephrine group will receive a continuous infusion containing epinephrine with a concentration of 0.02mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Interventions: Drug: Epinephrin
- Norepinephrine Group (Active Comparator): Patients in the norepinephrine group will receive a continuous infusion containing norepinephrine with a concentration of 0.02mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Interventions: Drug: Norepinephrine
- Phenylephrine Group (Active Comparator): Patients in the phenylephrine group will receive a continuous infusion containing phenylephrine with a concentration of 0.2mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Epinephrin — Patients in the epinephrine group will receive a continuous infusion containing epinephrine with a concentration of 0.02mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Arms: Epinephrine Group
Drug: Norepinephrine — Patients in the norepinephrine group will receive a continuous infusion containing norepinephrine with a concentration of 0.02mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Arms: Norepinephrine Group
Drug: Phenylephrine — Patients in the phenylephrine group will receive a continuous infusion containing phenylephrine with a concentration of 0.2mg/ml for intraoperative blood pressure management. The infusion will be started with 0.15mL/kg/h and will be titrated to receive a mean arterial pressure of at least 75mmHg.
  Arms: Phenylephrine Group

SUMMARY:
The use of catecholamines for blood pressure and hemodynamic management is essential during undergoing surgery. The type of the catecholamine with the most clinical meaningful effect is still unknown. Therefore, the investigators evaluate the effect of intraoperative continuous infusion of epinephrine, norepinephrine and phenylephrine on intraoperative cardiac output. The investigators further evaluate the effect of epinephrine, norepinephrine and phenylephrine on regional brain and regional tissue oxygenation during surgery.

DETAILED DESCRIPTION:
Background: The use of catecholamines for blood pressure and hemodynamic management is essential during undergoing surgery. The type of the catecholamine with the most clinical meaningful effect is still unknown. Therefore, the investigators evaluate the effect of intraoperative continuous infusion of epinephrine, norepinephrine and phenylephrine on intraoperative cardiac output. The investigators further evaluate the effect of epinephrine, norepinephrine and phenylephrine on regional brain and regional tissue oxygenation during surgery.

Methods: The study will include 225 patients ≥ 45 years of age undergoing moderate- to high-risk major open abdominal surgery lasting at least two hours in this prospective double-blinded randomized clinical trial. Patients will be randomly assigned to receive a continuous infusion of epinephrine, norepinephrine or phenylephrine for intraoperative blood pressure management. The primary outcome will be time weighted average (TWA) of cardiac output between continuous infusion of epinephrine, norepinephrine or phenylephrine. The secondary outcomes will be time weighted average of intraoperative brain regional oxygen saturation (brSO2) and tissue regional oxygen saturation (trSO2) between the groups.

Statistics: For the primary outcome, TWA of intraoperative cardiac output between the groups will be analyzed using an ANOVA. The primary outcome, TWA of intraoperative brSO2 and TWA of intraoperative trSO2 will be analysed using an ANOVA.

Level of originality: Data regarding the hemodynamic effects of commonly used intraoperative vasopressors on cardiac output are limited. In detail, effects of different types of catecholamines on hemodynamic parameters and subsequently tissue perfusion in the operative setting are lacking. This study will give further information of the different hemodynamic effects of the most used clinical used catecholamines which are used for intraoperative blood pressure management.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 45 years old
* Scheduled for moderate- to high-risk major open abdominal surgery expected to last at least two hours
* ASA physical status ≥ 2
* At least one of the following risk factors:

  1. Age ≥75years
  2. History of peripheral arterial disease
  3. History of coronary artery disease
  4. History of stroke or transient ischemic attack/Stroke
  5. History of chronic kidney disease
  6. Diabetes requiring medical treatment
  7. Current smoking or history of 15 pack-years
  8. History of heart failure
  9. Preoperative high-sensitivity Troponin T ≥14ng.L-1
  10. Preoperative NT-proBNP ≥200 pg.mL-1

Exclusion Criteria:

1. Scheduled for pheochromocytoma surgery
2. Scheduled for liver and kidney transplantation
3. Requiring preoperative intravenous vasopressor medications
4. Contraindications to epinephrine, norepinephrine or phenylephrine per clinical judgement
5. Permanent atrial fibrillation
6. Preoperative heart rate >110 bpm

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative cardiac output | Intraoperative
  Time weighted average of intraoperative cardiac output

SECONDARY OUTCOMES:
Secondary Outcome 1: Intraoperative brain regional oxygen saturation | Intraoperative
  Time weighted average of intraoperative brain regional oxygen saturation
Secondary Outcome 2: Intraoperative tissue regional oxygen saturation | Intraoperative
  Time weighted average of intraoperative tissue regional oxygen saturation

OTHER OUTCOMES:
Tertiary Outcome 1: NT-proBNP | Within the first three postoperative days
  Maximum concentration of NT-proBNP in the first three postoperative days
Tertiary Outcome 2: Troponin T | Within the first three postoperative days
  Maximum concentration of Troponin T in the first three postoperative days
Tertiary Outcome 3: Copeptin | Within the first three postoperative days
  Maximum concentration of Copeptin in the first three postoperative days
Exploratory Outcome 1: | Within the first three postoperative days
  Incidence of MINS
Exploratory Outcome 2: | Through study completion, on average 7 days
  Incidence of atrial fibrillation
Exploratory Outcome 3: | During hospitalization, on average 7 days
  Incidence of acute kidney injury
Exploratory Outcome 4: | During hospitalization, on average 7 days
  Incidence of myocardial infarction
Exploratory Outcome 5: | During hospitalization, on average 7 days
  Incidence of stroke
Exploratory Outcome 6: | During hospitalization, on average 7 days
  Incidence of wound related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No